CLINICAL TRIAL: NCT01959022
Title: A Pilot Study to Assess the Effects of Doxazosin on Polysomnography in PTSD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); Northern California Institute of Research and Education (Other)
Responsible Party: Principal Investigator, Anne Richards, Staff Psychiatrist, San Francisco Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-16907.5
Record Dates: First submitted 2013-10-04; First posted 2013-10-09 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Posttramatic Stress Disorder; Post-traumatic Stress Disorder; PTSD; Doxazosin; Nightmares; Sleep Disturbance
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Parasomnias | interventions — Doxazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxazosin XL (Experimental): Subjects will participate in a 2 week flexible-dose titration of doxazosin XL based on clinical response and adverse effects followed by 6 weeks of steady dose treatment.
  Interventions: Drug: Doxazosin XL

INTERVENTIONS:
Drug: Doxazosin XL — Subjects will participate in a 2 week flexible-dose titration of doxazosin based on clinical response and adverse effects followed by 6 weeks of steady dose treatment.
  Other Names: Cardura XL

SUMMARY:
This study will assess the effects of the medication doxazosin on sleep in men and women with PTSD. Sleep will be measured objectively at home using a portable sleep recorder and wrist actigraphy.

DETAILED DESCRIPTION:
This pilot study will assess the effects of doxazosin on objective measures of sleep in PTSD subjects using home ambulatory polysomnography. Twenty (20) men and women with chronic PTSD will be enrolled at the San Francisco Veterans Affairs Medical Center. After initial screening, subjects will complete 1 week of baseline assessments including 2 nights of home ambulatory polysomnography. They will then participate in a 2-week flexible-dose titration of doxazosin based on clinical response and adverse effects followed by 6 weeks of steady dose treatment ending with 2 nights of home polysomnography. Subjective and rater-based assessments will be conducted at baseline and at set intervals during and at the end of treatment. Wrist actigraphy measurements will also be made at baseline and at end of treatment as an economical, fairly valid and unobtrusive measure of sleep duration. We hypothesize that doxazosin will be associated with an increase in total sleep time (TST) and a decrease in wake time after sleep onset (WASO). We hypothesize that doxazosin will also be associated with clinical gains with respect to nightmares, subjective sleep quality, non-sleep PTSD symptoms, depression symptoms, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-69
2. Current full or partial syndromal PTSD of at least 3 months duration as indexed by the CAPS (Clinician-administered PTSD scale) score >30
3. CAPS recurrent distressing dreams item of >/= 5

Exclusion Criteria:

1. alcohol and or drug abuse/dependence in the last 3 months
2. lifetime history of any psychiatric disorder with psychotic features, bipolar disorder, obsessive-compulsive disorder
3. exposure to trauma within the last 3 months
4. prominent suicidal or homicidal ideation
5. sleep apnea diagnosis or positive screen for sleep apnea by Type III device.
6. neurologic disorder or systemic illness affecting CNS function
7. history of brain trauma or head injury with loss of consciousness greater than 10 minutes
8. chronic or unstable medical illness including unstable angina, myocardial infarction within the past 6 months, congestive heart failure, preexisting hypotension or orthostatic hypotension, chronic renal or hepatic failure, and pancreatitis
9. pregnancy, breastfeeding and/or refusal to use effective birth control
10. previous serious adverse reaction to an alpha-1-antagonist (such as priapism, hepatitis, angioedema, or intraoperative floppy iris syndrome)
11. current use of trazodone, hypnotics/benzodiazepines, mirtazapine, atypical antipsychotics, beta-adrenergic blockers, alpha-2-agonists, and current prazosin or other alpha-1-antagonists
12. previous non-response to prazosin for treatment of PTSD related sleep disturbance

Participants taking SSRIs, bupropion, venlafaxine and duloxetine may be included if they have been on a stable dose for 2 months. Participants may be included if they have been stable in psychotherapy treatment for 2 months and/or if they begin no new psychotherapy while in the trial.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in mean total sleep time and wake-time after sleep onset as measured by polysomnography and actigraphy | baseline and 8 weeks
Change in REM sleep time and REM period duration as measured by polysomnography | baseline and 8 weeks

SECONDARY OUTCOMES:
Change in mean scores on the CAPS, CAPS sleep and distressing dreams items, PCL, BDI, ISI, PSQI, PSQI-A and QOLI | baseline and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne Richards, MD, MPH, Principal Investigator — San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] De Jong J, Wauben P, Huijbrechts I, Oolders H, Haffmans J. Doxazosin treatment for posttraumatic stress disorder. J Clin Psychopharmacol. 2010 Feb;30(1):84-5. doi: 10.1097/JCP.0b013e3181c827ae. No abstract available. PMID 20075659
- [Background] Taylor FB, Martin P, Thompson C, Williams J, Mellman TA, Gross C, Peskind ER, Raskind MA. Prazosin effects on objective sleep measures and clinical symptoms in civilian trauma posttraumatic stress disorder: a placebo-controlled study. Biol Psychiatry. 2008 Mar 15;63(6):629-32. doi: 10.1016/j.biopsych.2007.07.001. Epub 2007 Sep 14. PMID 17868655